CLINICAL TRIAL: NCT02750774
Title: A Customized Low Glycaemic-index (GI) Diet, Introduced at First Trimester of Pregnancy by Both Gynecologist and Dietitian, Prevents Large for Gestational Age (LGA) Newborns in Overweight/Obese Pregnant Women
Brief Title: An Early-customized Low Glycaemic-index (GI) Diet Prevents LGA Babies in Overweight/Obese Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Dr. Elisabetta Petrella (Unknown)
Responsible Party: Principal Investigator, Prof. Facchinetti Fabio, Professor Fabio Facchinetti, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pratica CE 136/15
Record Dates: First submitted 2016-04-14; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Maternal Obesity Complicating Pregnancy, Birth,or Puerperium; Gestational Diabetes Mellitus; Birthweight; Large for Gestational Age (LGA); Caloric Restriction; Lifestyle Intervention
MeSH Terms: conditions — Diabetes, Gestational; Birth Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Glycemic Index Group (Experimental): Women in the low- glycaemic index group received a dietary intervention based on 3 main meals and 3 snacks, with a precise macronutrient composition, and a physical activity counseling according to the ACOG and ACSM recommendations.
  Interventions: Behavioral: Low-glycemic index group
- Standard Care Group (Other): Women in the Standard Care Group received a simple nutritional booklet regarding lifestyle, which was in agreement with the Italian Guidelines for a healthy diet during pregnancy that included general advice regarding food consumption and physical activity.
  Interventions: Other: Standard Care Group

INTERVENTIONS:
Behavioral: Low-glycemic index group — The dietary intervention consisted of the prescription of a Mediterranean style, low-glycaemic, low-fat, exchange diet (3 main meals and 3 snacks) with a total intake of 1500 kcal/day. In light of the PA, the dietitian adds 200 kcal/day for obese, 300 kcal/day for overweight women. The diet had a target macronutrient composition of 55% carbohydrates (80% complex carbohydrates with a low glycaemic index and 20% simple carbohydrates), 20% protein (50% animal and 50% vegetable) and 25% fat (12% mono-unsaturated, 7% polyunsaturated and 6% saturated) with moderately low saturated fat levels. The daily intake of carbohydrates was at least 225 g/day. The exercise intervention was focused on developing a more active lifestyle. The PA prescription is consistent with recommendations by the ACOG and ACSM for pregnant women. The "talk test" (being able to maintain a conversation during activity) was suggested to monitor the exercise intensity.
  Arms: Low-Glycemic Index Group
Other: Standard Care Group — Women randomized to the Standard Care Group received general information about healthy lifestyle during pregnancy, according to the Guidelines
  Arms: Standard Care Group

SUMMARY:
High pre-pregnancy body mass index (BMI) and excessive gestational weight gain (GWG) are associated with many unfavourable maternal and neonatal outcomes.

Adherence to lifestyle recommendations could be a major determinant of the efficacy on preventing unfavorable outcomes, namely among overweight/obese women. Previous studies investigated adherence to specific dietary patterns and their effect on pregnancy outcomes; however, no study has investigated adherence among overweight/obese pregnant women and its effect on the onset of several maternal-neonatal outcomes.

This study aimed to determine whether the prescription of a lifestyle program, consisting of a customized low-glycemic index (GI) diet and a physical activity program, in overweight and obese women could affect the occurrence LGA babies. It also aimed to determine whether this kind of prescription influences the adherence to healthier eating habits, and how this, in turn, can influence the occurrence LGA.

DETAILED DESCRIPTION:
High pre-pregnancy BMI and excessive GWG are associated with many unfavourable maternal and neonatal outcomes and are independent risk factors for gestational diabetes mellitus (GDM) and large for gestatiola age (LGA) babies. Overweight/obese women should be counselled regarding their body weight before conception; however, most women have access to obstetricians only when they are pregnant. The Institute of Medicine (IOM) revised the guidelines of recommended GWG according to the BMI; however, only a minority of women succeed in reaching the recommended GWG. Among the interventions aimed at preventing excessive GWG, few have demonstrated efficacy in high-risk populations; the principal issues are population heterogeneity, the interventional methods, and the timing of the interventional programs. Additionally, lifestyle interventions did not have a substantial effect on other clinical outcomes. Dietary advice to prevent gestational diabetes mellitus (GDM) appears to be beneficial in general, although the results are overly heterogeneous. A systematic review concerning exercise alone demonstrated no effect on preventing GDM, whereas another study showed only a slight protective effect. The reports evaluating the efficacy of diverse approaches (exercise, diet, lifestyle interventions, dietary supplements) to prevent GDM are of poor quality. Adherence to lifestyle recommendations could be a major determinant of their efficacy, specifically among overweight/obese women. Previous studies investigated adherence to specific dietary patterns and their effect on pregnancy outcomes; however, no study has investigated adherence among overweight/obese pregnant women and its effect on the onset of GDM. Nowadays, there are insufficient evidences for recommend a specific diet in preventing LGA babies.

This study aimed to determine whether the prescription of an early lifestyle program, consisting of a low-glycemic index (GI) caloric restriction and physical activity (PA), in overweight and obese women could affect the occurrence of LGA newborns. It also aimed to determine whether this kind of prescription influences the adherence to healthier eating habits, and how this, in turn, can influence the occurrence of LGA babies.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* singleton pregnancy
* BMI >= 25 kg/m2

Exclusion Criteria:

* Chronic diseases including diabetes mellitus (first trimester glycosuria> 100 mg/dl or fasting plasma glucose ≥126 mg/dL or random glycemia ≥ 200 mg/dL) and hypertension
* Previous GDM
* Medical conditions or dietary supplements that might affect the body weight (i.e., thyroid diseases)
* Previous bariatric surgery
* Smoking habits
* Contraindications to exercise
* Intent to deliver outside our hospital

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Large-for-gestational-age (LGA) occurrence | At delivery
  LGA babies were defined if birthweight centile was ≥ 90°, and it was measured at delivery
Gestational Diabetes Mellitus (GDM) occurrence | At 24-26 weeks
  The diagnosis of GDM was made for any glucose value exceeding the normal cut-off, according to the Guidelines

SECONDARY OUTCOMES:
Gestational Weight Gain (GWG) | At baseline, at 16, 20, 28 and 36 weeks, at delivery and 3 months after delivery
  Excessive GWG is related to unfavorable pregnancy outcomes. Weight gain is measured at each follow-up visit, at delivery and 3 months after delivery in both groups, to evaluate possible effects of the intervention.
Pre-term Birth (PTB) | At delivery
  Both spontaneous and medically indicated preterm births are associated with obesity. We recorded cases of preterm birth, if it was spontaneous or not and the eventual indication.
Neonatal hypoglycemia | Within 24 hours after delivery
  Altered maternal glucose metabolism is associated with neonatal hypoglicemia
Neonatal Intensive Care Unit (NICU) admission | Within 24 hours after delivery
  Maternal overweight and obesity are related to higher prevalence of neonatal complications

CONTACTS AND LOCATIONS:
Locations (1):
- Mother-Infant Department, University of Modena and Reggio Emilia, Italy, Modena, Italy

IPD SHARING:
Plan to Share IPD: Yes